CLINICAL TRIAL: NCT02487771
Title: Kansas University DHA Outcome Study (KUDOS) Follow-Up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Susan Carlson, PhD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Susan Carlson, PhD, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11406; 1R01HD047315 (NIH)
Record Dates: First submitted 2012-06-18; First posted 2015-07-01 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy
Keywords: DHA; childhood development
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Capsule (Placebo Comparator)
  Interventions: Drug: Placebo Capsule
- DHA Capsule (Experimental)
  Interventions: Drug: DHA

INTERVENTIONS:
Drug: DHA — 600 mg DHA capsule
  Other Names: docosahexaenoic acid
  Arms: DHA Capsule
Drug: Placebo Capsule — 600 mg of Soybean Oil and Corn Oil, which does not contain any DHA
  Arms: Placebo Capsule

SUMMARY:
This is a continuation study to KUDOS (NCT00266825). The purpose of this study is to follow-up with participants on the original study to determine if the effects of increasing DHA intake during pregnancy increase cognitive development in 2 to 6 year-old children.

DETAILED DESCRIPTION:
Numerous trials show benefits of postnatal DHA supplementation for visual acuity. There are also numerous observational(not intervention)studies that link higher maternal DHA status during pregnancy to higher cognitive function. Intervention studies that increase DHA exposure during fetal life and that measure cognitive development of infants are lacking; and no study to date has systematically followed children whose mothers were randomly assigned to DHA supplementation to school age with regular 6 month assessments of age-appropriate assessments of cognitive development. The absence of such studies is a serious limitation because there is evidence that differences in cognitive function due to such interventions do not become robust until around age 4 years. Women in the US consume low amounts of DHA compared to other world populations, and this likely means less DHA transfer to the fetus than in many other populations. Prenatal DHA exposure may be more important than postnatal exposure, because animal studies show critical windows for brain DHA accumulation in relation to effects on neurotransmitters such as serotonin, dopamine and GABA.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females 16.0-35.0 years of age (inclusive) at 8-20 weeks gestation at enrollment (date/ultrasound)
* Agree to consume study capsules from enrollment until delivery
* Agree to return to the study center for delivery
* BMI < 40
* No serious illnesses (e.g., cancer, diabetes, lupus, hepatitis, sexually transmitted diseases, not HIV positive)
* Available by telephone

Exclusion Criteria:

* Less than 16 or greater than 35 years of age
* BMI < 40
* Serious illness such as cancer, lupus, hepatitis, sexually transmitted disease or HIV positive
* Expecting multiple infants
* Diabetes or gestational diabetes at baseline
* Elevated blood pressure due to any cause
* Not planning to return to the study center for delivery
* Gestational age at baseline < 8 weeks or >20 weeks
* Unable or unwilling to agree to consume capsules until delivery
* Unable to provide informed consent in English

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 190 (Actual)
Dates: Start 2008-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Carlson, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Colombo J, Shaddy DJ, Gustafson K, Gajewski BJ, Thodosoff JM, Kerling E, Carlson SE. The Kansas University DHA Outcomes Study (KUDOS) clinical trial: long-term behavioral follow-up of the effects of prenatal DHA supplementation. Am J Clin Nutr. 2019 May 1;109(5):1380-1392. doi: 10.1093/ajcn/nqz018. PMID 31004139
- [Derived] Kerling EH, Hilton JM, Thodosoff JM, Wick J, Colombo J, Carlson SE. Effect of Prenatal Docosahexaenoic Acid Supplementation on Blood Pressure in Children With Overweight Condition or Obesity: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2019 Feb 1;2(2):e190088. doi: 10.1001/jamanetworkopen.2019.0088. PMID 30794304
- See also: Main KUDOS Study Posting on Clinicaltrials.gov — http://clinicaltrials.gov/ct2/show/NCT00266825

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 7/17/2008 to 4/24/2012.
Pre-assignment Details: Participants were required to have been enrolled in the parent trial.
Period: Overall Study
Arm/Group | Placebo Capsule | DHA Capsule
Started | 91 | 99
Completed | 81 | 85
Not Completed | 10 | 14
Not completed — Lost to Follow-up | 2 | 3
Not completed — Moved out of area | 5 | 6
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Population: Families who completed the parent trial were offered enrollment when their child was 2 yrs of age.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Capsule | DHA Capsule | Total
Number analyzed (Participants) | 91 | 99 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.01 (0.03) | 2.01 (0.03) | 2.01 (0.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 55 | 95
  Male | 51 | 44 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 10 | 9 | 19
  Not Hispanic | 81 | 90 | 171
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 33 | 33 | 66
  Not Black | 58 | 66 | 124
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91 | 99 | 190

OUTCOME MEASURES:

1. Primary Outcome: Weschler Preschool and Primary Scale of Intelligence, 3rd Edition; Full Scale IQ
Description: The Full Scale IQ score from the Weschler Preschool and Primary Scale of Intelligence, 3rd Edition is a standardized measure of a child's general intellectual ability based upon assessments of verbal, cognitive, and performance domains. At three years the Full Scale IQ score has a range of 41 (poorest performance) to 155 (best performance). For the older ages the score can range from 40 to 160. For all ages the assessment is normed to a Mean = 100, St Dev = 15.
Time Frame: 36 Months
Population: Missing data for participants dues to attrition, missed appointments, refusals, or questionable test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 74 | 88
units on a scale | 98.78 (15.43) | 98.75 (15.75)

2. Primary Outcome: Weschler Preschool and Primary Scale of Intelligence, 3rd Edition; Full Scale IQ
Description: as for outcome 1
Time Frame: 48 Months
Population: Missing data for participants dues to attrition, missed appointments, refusals, or questionable test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 66 | 79
units on a scale | 97.52 (15.32) | 99.72 (16.10)

3. Primary Outcome: Weschler Preschool and Primary Scale of Intelligence, 3rd Edition; Full Scale IQ
Description: as for outcome 1
Time Frame: 72 Months
Population: Missing data for participants dues to attrition, missed appointments, refusals, or questionable test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 69 | 81
units on a scale | 100.67 (14.70) | 102.21 (14.02)

4. Primary Outcome: Cognitive Function Score - Peabody Picture Vocabulary Test
Description: The Peabody Picture Vocabulary Test, 3rd Edition provides a standardized assessment of a person's receptive vocabulary. The Standard Score can range from 40 (poorest performance) to 160 (best performance) and has been normed to a Mean = 100, St Dev = 15.
Time Frame: 60 Months
Population: Missing data due to attrition, missed appointments, refusals, or questionable test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 74 | 85
units on a scale | 101.07 (14.92) | 102.35 (15.33)

5. Primary Outcome: Cognitive Function Score - Test of Preschool Early Literacy
Description: The Test of Preschool Early Literacy provides a standardized Early Literacy Index score, a measure of general, early literacy skills that relate to later reading and writing skill acquisition. The score is based on assessments of vocabulary, print knowledge, and phonological awareness. The score can range from 40 (poorest performance) to 144 (best performance) and has been normed to a Mean = 100, St Dev = 15.
Time Frame: 42 Months
Population: Missing data due to attrition, missed appointments, refusals, or questionable test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 71 | 87
units on a scale | 92.99 (18.76) | 95.08 (18.80)

6. Primary Outcome: Weschler Preschool and Primary Scale of Intelligence, 3rd Edition; Verbal IQ
Description: The Verbal IQ score from the Weschler Preschool and Primary Scale of Intelligence, 3rd Edition is a standardized measure of a child's verbal ability based upon assessments of vocabulary, general knowledge, and reasoning. At three years the Verbal IQ score has a range of 49 (poorest performance) to 150 (best performance). For the older ages the score can range from 46 to 155. For all ages the assessment is normed to a Mean = 100, St Dev = 15.
Time Frame: 36 Months
Population: Missing data due to attrition, missed appointments, refusals, or questionable test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 77 | 91
units on a scale | 100.98 (14.22) | 101.10 (16.51)

7. Primary Outcome: Weschler Preschool and Primary Scale of Intelligence, 3rd Edition; Verbal IQ
Description: as for outcome 6
Time Frame: 48 Months
Population: Missing data due to attrition, missed appointments, refusals, or questionable test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 67 | 80
units on a scale | 99.30 (15.31) | 100.13 (16.13)

8. Primary Outcome: Weschler Preschool and Primary Scale of Intelligence, 3rd Edition; Verbal IQ
Description: as for outcome 6
Time Frame: 72 Months
Population: Missing data due to attrition, missed appointments, refusals, or questionable test
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 70 | 81
units on a scale | 101.53 (14.20) | 102.44 (14.88)

9. Secondary Outcome: Adaptive Regulation Assessment
Description: The Parent Rating Scales of the Behavior Assessment System for Children 2nd Edition measures different aspects of a child's behaviors as reported by a parent. Externalizing Problems is a measure of Aggression and Hyperactivity. Internalizing Problems is a measure of Anxiety, Depression, and Somatization. The Behavioral Symptoms Index is a more global measure of behavior problems and combines Externalizing Problems with the measure of Depression from Internalizing Problems, and additional measures of Atypicality, Withdrawal, and Attention Problems. Adaptive Skills is a measure of Adaptability, Social Skills, Activities of Daily Living, Functional Communication, and at age 6 years Leadership. All scores are derived from the general, combined sex normative tables of T-Scores. For Adaptive Skills higher T-Scores reflect a more optimal outcome. For all other measures lower T-Scores reflect a more optimal outcome. All T-Scores were standardized with a Mean = 50, St Dev = 10.
Time Frame: 36 Months
Population: Missing data due to attrition, missed appointments, refusals.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 71 | 82
T-scores
  Externalizing Problems | 48.17 (6.86) | 49.11 (7.85)
  Internalizing Problems | 49.31 (9.67) | 49.10 (8.05)
  Behavioral Symptoms | 47.99 (7.13) | 49.46 (6.85)
  Adaptive Skills | 54.00 (7.49) | 52.56 (7.23)

10. Secondary Outcome: Adaptive Regulation Assessment
Description: as for outcome 9
Time Frame: 48 Months
Population: Missing data due to attrition, missed appointments, refusals.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 74 | 85
T-scores
  Externalizing Problems | 48.87 (8.22) | 50.08 (8.22)
  Internalizing Problems | 47.30 (8.65) | 47.46 (8.73)
  Behavioral Symptoms | 49.42 (8.62) | 50.59 (7.20)
  Adaptive Skills | 50.15 (8.76) | 47.72 (8.40)

11. Secondary Outcome: Adaptive Regulation Assessment
Description: as for outcome 9
Time Frame: 60 Months
Population: Missing data due to attrition, missed appointments, refusals.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 72 | 83
T-scores
  Externalizing Problems | 48.94 (8.71) | 50.43 (9.22)
  Internalizing Problems | 49.99 (7.96) | 49.21 (8.75)
  Behavioral Symptoms | 50.17 (7.66) | 50.78 (8.19)
  Adaptive Skills | 52.09 (8.18) | 50.96 (8.13)

12. Secondary Outcome: Adaptive Regulation Assessment
Description: as for outcome 9
Time Frame: 72 Months
Population: Missing data due to attrition, missed appointments, refusals.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 67 | 75
T-scores
  Externalizing Problems | 50.10 (9.68) | 49.37 (6.76)
  Internalizing Problems | 46.80 (7.80) | 45.96 (8.35)
  Behavioral Symptoms | 48.99 (8.09) | 49.17 (6.72)
  Adaptive Skills | 51.80 (8.09) | 49.73 (9.77)

13. Other Pre Specified Outcome: Anthropometrics: Weight-for-age
Description: Biannually child weight was measured one time standing without shoes and in the lightest layer of clothing to the nearest 0.1 kg on an electronic scale (Cardinal Detecto 8430, Webb City, MS, USA).
Time Frame: 2 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 85 | 97
Kilogram (kg) | 12.66 (1.51) | 12.99 (1.44)

14. Other Pre Specified Outcome: Anthropometrics: Weight-for-age
Description: as for outcome 13
Time Frame: 2.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 86 | 97
Kilogram (kg) | 13.70 (1.66) | 14.08 (1.51)

15. Other Pre Specified Outcome: Anthropometrics: Weight-for-age
Description: as for outcome 13
Time Frame: 3 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 87 | 97
Kilogram (kg) | 14.83 (1.76) | 15.16 (1.60)

16. Other Pre Specified Outcome: Anthropometrics: Height-for-Age
Description: Biannually child stature was measured one time standing without shoes and in the lightest layer of clothing to the nearest 0.1 cm using a wall mounted statiometer (Health O Meter® Professional, McCook IL, USA). Braids, ponytails or other hair artifacts were removed or subtracted when needed.
Time Frame: 2 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 83 | 97
Centimeters (cm) | 85.91 (3.42) | 86.54 (3.09)

17. Other Pre Specified Outcome: Anthropometrics: Weight-for-age
Description: as for outcome 13
Time Frame: 3.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 85 | 95
Kilogram (kg) | 15.90 (1.91) | 16.36 (1.85)

18. Other Pre Specified Outcome: Anthropometrics: Weight-for-age
Description: as for outcome 13
Time Frame: 4 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 87 | 91
Kilogram (kg) | 17.13 (2.11) | 17.71 (2.10)

19. Other Pre Specified Outcome: Anthropometrics: Weight-for-age
Description: as for outcome 13
Time Frame: 4.5 years
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 86 | 91
Kilogram (kg) | 18.29 (2.38) | 18.96 (2.55)

20. Other Pre Specified Outcome: Anthropometrics: Weight-for-age
Description: as for outcome 13
Time Frame: 5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 83 | 88
Kilogram (kg) | 19.75 (2.85) | 20.33 (3.05)

21. Other Pre Specified Outcome: Anthropometrics: Weight-for-age
Description: as for outcome 13
Time Frame: 5.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 85
Kilogram (kg) | 21.23 (3.5) | 21.73 (3.18)

22. Other Pre Specified Outcome: Anthropometrics: Weight-for-age
Description: as for outcome 13
Time Frame: 6 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 85
Kilogram (kg) | 22.68 (4.16) | 23.14 (3.66)

23. Other Pre Specified Outcome: Anthropometrics: Height-for-Age
Description: as for outcome 16
Time Frame: 2.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 86 | 96
Centimeters (cm) | 90.66 (3.10) | 91.17 (3.69)

24. Other Pre Specified Outcome: Anthropometrics: Height-for-Age
Description: as for outcome 16
Time Frame: 3 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 87 | 96
Centimeters (cm) | 94.90 (3.48) | 95.29 (3.52)

25. Other Pre Specified Outcome: Anthropometrics: Height-for-Age
Description: as for outcome 16
Time Frame: 3.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 85 | 95
Centimeters (cm) | 98.96 (3.79) | 99.27 (3.58)

26. Other Pre Specified Outcome: Anthropometrics: Height-for-Age
Description: as for outcome 16
Time Frame: 4 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 87 | 91
Centimeters (cm) | 102.77 (3.82) | 103.32 (3.91)

27. Other Pre Specified Outcome: Anthropometrics: Height-for-Age
Description: as for outcome 16
Time Frame: 4.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 86 | 91
Centimeters (cm) | 106.39 (4.23) | 107.11 (4.09)

28. Other Pre Specified Outcome: Anthropometrics: Height-for-Age
Description: as for outcome 16
Time Frame: 5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 83 | 88
Centimeters (cm) | 110.03 (4.30) | 110.58 (4.23)

29. Other Pre Specified Outcome: Anthropometrics: Height-for-Age
Description: as for outcome 16
Time Frame: 5.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 85
Centimeters (cm) | 113.41 (4.39) | 114.01 (4.34)

30. Other Pre Specified Outcome: Anthropometrics: Height-for-Age
Description: as for outcome 16
Time Frame: 6 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 85
Centimeters (cm) | 116.76 (4.74) | 117.22 (4.60)

31. Other Pre Specified Outcome: Anthropometrics: Body Mass Index-for-age
Description: Biannually child body mass index (BMI) was calculated using the standard equation: BMI = kg/m^2.
Time Frame: 2 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Body mass index (kg/m^2)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 83 | 97
Body mass index (kg/m^2) | 17.13 (1.53) | 17.31 (1.28)

32. Other Pre Specified Outcome: Anthropometrics: Body Mass Index-for-age
Description: Biannually child body mass index (BMI) was calculated using the standard equation: BMI = kg/m^2.
Time Frame: 2.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Body mass index (kg/m2)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 85 | 94
Body mass index (kg/m2) | 16.65 (1.37) | 16.92 (1.27)

33. Other Pre Specified Outcome: Anthropometrics: Body Mass Index-for-age
Description: Biannually child body mass index (BMI) was calculated using the standard equation: BMI = kg/m^2.
Time Frame: 3 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Body mass index (kg/m2)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 87 | 96
Body mass index (kg/m2) | 16.44 (1.33) | 16.67 (1.25)

34. Other Pre Specified Outcome: Anthropometrics: Body Mass Index-for-age
Description: Biannually child body mass index (BMI) was calculated using the standard equation: BMI = kg/m^2.
Time Frame: 3.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Body mass index (kg/m2)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 85 | 95
Body mass index (kg/m2) | 16.21 (1.36) | 16.57 (1.32)

35. Other Pre Specified Outcome: Anthropometrics: Body Mass Index-for-age
Description: Biannually child body mass index (BMI) was calculated using the standard equation: BMI = kg/m^2.
Time Frame: 4 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Body mass index (kg/m2)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 87 | 91
Body mass index (kg/m2) | 16.18 (1.38) | 16.56 (1.46)

36. Other Pre Specified Outcome: Anthropometrics: Body Mass Index-for-age
Description: Biannually child body mass index (BMI) was calculated using the standard equation: BMI = kg/m^2.
Time Frame: 4.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Body mass index (kg/m2)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 86 | 91
Body mass index (kg/m2) | 16.12 (1.51) | 16.49 (1.74)

37. Other Pre Specified Outcome: Anthropometrics: Body Mass Index-for-age
Description: Biannually child body mass index (BMI) was calculated using the standard equation: BMI = kg/m^2.
Time Frame: 5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Body mass index (kg/m2)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 83 | 88
Body mass index (kg/m2) | 16.27 (1.83) | 16.58 (1.97)

38. Other Pre Specified Outcome: Anthropometrics: Body Mass Index-for-age
Description: Biannually child body mass index (BMI) was calculated using the standard equation: BMI = kg/m^2.
Time Frame: 5.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Body mass index (kg/m2)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 85
Body mass index (kg/m2) | 16.46 (2.22) | 16.68 (1.95)

39. Other Pre Specified Outcome: Anthropometrics: Body Mass Index-for-age
Description: Biannually child body mass index (BMI) was calculated using the standard equation: BMI = kg/m^2.
Time Frame: 6 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Body mass index (kg/m2)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 85
Body mass index (kg/m2) | 16.57 (2.51) | 16.81 (2.27)

40. Other Pre Specified Outcome: Anthropometrics: Head Circumference-for-age
Description: Biannually child head circumference was measured to the nearest 0.1 cm using standard technique (tape positioned just above the eyebrows, above the ears and around the biggest part of the back of the head; tape pulled snuggly to compress hair and underlying soft tissue). Braids, ponytails, glasses or other artifacts were removed whenever possible.
Time Frame: 2 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 94
Centimeters (cm) | 48.40 (1.29) | 48.50 (1.38)

41. Other Pre Specified Outcome: Anthropometrics: Head Circumference-for-age
Description: as for outcome 40
Time Frame: 2.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 85 | 95
Centimeters (cm) | 49.18 (1.36) | 49.21 (1.37)

42. Other Pre Specified Outcome: Anthropometrics: Head Circumference-for-age
Description: as for outcome 40
Time Frame: 3 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 87 | 97
Centimeters (cm) | 49.64 (1.34) | 49.75 (1.34)

43. Other Pre Specified Outcome: Anthropometrics: Head Circumference-for-age
Description: as for outcome 40
Time Frame: 3.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 84 | 95
Centimeters (cm) | 50.05 (1.35) | 50.15 (1.28)

44. Other Pre Specified Outcome: Anthropometrics: Head Circumference-for-age
Description: as for outcome 40
Time Frame: 4 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 86 | 91
Centimeters (cm) | 50.47 (1.37) | 50.62 (1.33)

45. Other Pre Specified Outcome: Anthropometrics: Head Circumference-for-age
Description: as for outcome 40
Time Frame: 4.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 86 | 91
Centimeters (cm) | 50.78 (1.36) | 50.95 (1.42)

46. Other Pre Specified Outcome: Anthropometrics: Head Circumference-for-age
Description: as for outcome 40
Time Frame: 5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 83 | 88
Centimeters (cm) | 51.04 (1.48) | 51.37 (1.48)

47. Other Pre Specified Outcome: Anthropometrics: Head Circumference-for-age
Description: as for outcome 40
Time Frame: 5.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 84
Centimeters (cm) | 51.48 (1.42) | 51.58 (1.42)

48. Other Pre Specified Outcome: Anthropometrics: Head Circumference-for-age
Description: as for outcome 40
Time Frame: 6 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 80 | 84
Centimeters (cm) | 51.77 (1.51) | 51.93 (1.59)

49. Other Pre Specified Outcome: Dietary Intake
Description: Biannually a registered dietitian assessed child diet by a standardized 24 hour dietary recall with three-pass approach. When necessary both the parent and child participated in the recall process to increase overall reliability. Recalls were entered into Nutrition Data System for Research (NDS-R versions 2006-2016, University of Minnesota, Minneapolis, MN, USA) and were checked for accuracy by a second dietitian. Reliability and caloric intake data are presented here. Reliability is defined as the dietitian's subjective assessment of the family's ability to recall the majority of food items consumed during the 24 hour period and within reasonable serving sizes. Caloric intake is the mean kcal per day from reliable recalls only.
Time Frame: 2 years
Population: Missing data due to attrition, missed appointments, refusals or questionable intake
Measure: Mean (Standard Deviation); unit: kilocalorie
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 76 | 88
kilocalorie | 1226 (384) | 1210 (439)

50. Other Pre Specified Outcome: Dietary Intake
Description: as for outcome 49
Time Frame: 2.5 years
Population: Missing data due to attrition, missed appointments, refusals or questionable intake
Measure: Mean (Standard Deviation); unit: kilocalorie
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 75 | 88
kilocalorie | 1256 (413) | 1234 (396)

51. Other Pre Specified Outcome: Dietary Intake
Description: as for outcome 49
Time Frame: 3 years
Population: Missing data due to attrition, missed appointments, refusals or questionable intake
Measure: Mean (Standard Deviation); unit: kilocalorie
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 74 | 90
kilocalorie | 1364 (418) | 1285 (415)

52. Other Pre Specified Outcome: Dietary Intake
Description: as for outcome 49
Time Frame: 3.5 years
Population: Missing data due to attrition, missed appointments, refusals or questionable intake
Measure: Mean (Standard Deviation); unit: kilocalorie
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 77 | 86
kilocalorie | 1340 (361) | 1275 (407)

53. Other Pre Specified Outcome: Dietary Intake
Description: as for outcome 49
Time Frame: 4 years
Population: Missing data due to attrition, missed appointments, refusals or questionable intake
Measure: Mean (Standard Deviation); unit: kilocalorie
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 76 | 82
kilocalorie | 1468 (472) | 1388 (398)

54. Other Pre Specified Outcome: Dietary Intake
Description: as for outcome 49
Time Frame: 4.5 years
Population: Missing data due to attrition, missed appointments, refusals or questionable intake
Measure: Mean (Standard Deviation); unit: kilocalorie
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 79 | 84
kilocalorie | 1459 (439) | 1432 (423)

55. Other Pre Specified Outcome: Dietary Intake
Description: as for outcome 49
Time Frame: 5 years
Population: Missing data due to attrition, missed appointments, refusals or questionable intake
Measure: Mean (Standard Deviation); unit: kilocalorie
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 73 | 75
kilocalorie | 1412 (380) | 1466 (479)

56. Other Pre Specified Outcome: Dietary Intake
Description: as for outcome 49
Time Frame: 5.5 years
Population: Missing data due to attrition, missed appointments, refusals or questionable intake
Measure: Mean (Standard Deviation); unit: kilocalorie
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 64 | 73
kilocalorie | 1557 (436) | 1532 (458)

57. Other Pre Specified Outcome: Dietary Intake
Description: as for outcome 49
Time Frame: 6 years
Population: Missing data due to attrition, missed appointments, refusals or questionable intake
Measure: Mean (Standard Deviation); unit: kilocalorie
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 70 | 73
kilocalorie | 1655 (487) | 1495 (469)

58. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Biannually child blood pressure was measured in triplicate using an automatic pressure cuff (GE Carescape V100, Chicago, IL, USA) while children were seated in a resting state. Raw averages are reported here, including outliers. Not all subjects participated in triplicate measures.
Time Frame: 4 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 78 | 86
Millimeters of mercury (mmHg) | 100.0 (10.8) | 98.7 (8.3)

59. Other Pre Specified Outcome: Systolic Blood Pressure
Description: as for outcome 58
Time Frame: 4.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 85
Millimeters of mercury (mmHg) | 101.0 (8.7) | 100.3 (7.6)

60. Other Pre Specified Outcome: Systolic Blood Pressure
Description: as for outcome 58
Time Frame: 5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 78 | 83
Millimeters of mercury (mmHg) | 99.5 (7.1) | 98.2 (8.3)

61. Other Pre Specified Outcome: Systolic Blood Pressure
Description: as for outcome 58
Time Frame: 5.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 77 | 84
Millimeters of mercury (mmHg) | 102.1 (8.1) | 103.5 (9.1)

62. Other Pre Specified Outcome: Systolic Blood Pressure
Description: as for outcome 58
Time Frame: 6 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 76 | 83
Millimeters of mercury (mmHg) | 99.6 (8.1) | 98.9 (7.7)

63. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: as for outcome 58
Time Frame: 4 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 78 | 86
Millimeters of mercury (mmHg) | 62.1 (11.2) | 58.8 (7.7)

64. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: as for outcome 58
Time Frame: 4.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 85
Millimeters of mercury (mmHg) | 63.3 (9.5) | 61.0 (6.8)

65. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: as for outcome 58
Time Frame: 5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 78 | 83
Millimeters of mercury (mmHg) | 58.9 (5.9) | 58.3 (7.7)

66. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: as for outcome 58
Time Frame: 5.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 77 | 84
Millimeters of mercury (mmHg) | 62.5 (8.0) | 61.5 (7.6)

67. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: as for outcome 58
Time Frame: 6 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 76 | 83
Millimeters of mercury (mmHg) | 60.1 (6.1) | 59.0 (5.3)

68. Other Pre Specified Outcome: Heart Rate
Description: Biannually child heart rate was measured in triplicate using an automatic pressure cuff (GE Carescape V100, Chicago, IL, USA) while children were seated in a resting state. Raw averages are reported here, including outliers. Not all subjects participated in triplicate measures.
Time Frame: 4 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 78 | 86
Beats per minute (BPM) | 92.6 (9.9) | 93.1 (12.0)

69. Post Hoc Outcome: Anthropometrics: Body Composition
Description: Child body composition was measured between 5 and 6 years of age by BOD POD air displacement plethysmography (COSMED, Concord, CA, USA). Methods adhered to standard testing protocol (tight-fitting one-piece swimsuit and swim cap, duplicate or triplicate measure of body volume and predicted thoracic gas volume). Fat and fat free mass to the nearest 0.1 kg are presented as means with standard deviations. Normative data are not available in this pediatric population.
Time Frame: 5 to 5.5 years old
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 76 | 78
Kilogram (kg)
  Fat Mass | 4.89 (1.59) | 5.17 (1.66)
  Fat Free Mass | 14.60 (2.31) | 15.18 (2.10)

70. Other Pre Specified Outcome: Heart Rate
Description: as for outcome 68
Time Frame: 4.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 81 | 85
Beats per minute (BPM) | 91.1 (10.7) | 91.1 (9.0)

71. Other Pre Specified Outcome: Heart Rate
Description: as for outcome 68
Time Frame: 5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 78 | 83
Beats per minute (BPM) | 90.4 (10.7) | 90.4 (9.6)

72. Other Pre Specified Outcome: Heart Rate
Description: as for outcome 68
Time Frame: 5.5 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 77 | 84
Beats per minute (BPM) | 87.9 (12.4) | 87.2 (11.0)

73. Other Pre Specified Outcome: Heart Rate
Description: as for outcome 68
Time Frame: 6 years
Population: Missing data due to attrition, missed appointments or refusals
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Placebo Capsule | DHA Capsule
Number analyzed (Participants) | 76 | 83
Beats per minute (BPM) | 84.2 (11) | 85.4 (10.8)

ADVERSE EVENTS:
Description: Adverse events were not analyzed as part of this follow up.
Arm/Group | Placebo Capsule | DHA Capsule
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes